CLINICAL TRIAL: NCT07189247
Title: Evaluation of Fibromyalgia Frequency and Pain Parameters in Women With Polycystic Ovary Syndrome: A Prospective Single-Blind Study
Brief Title: Evaluation of Fibromyalgia Frequency and Pain Parameters in Women With Polycystic Ovary Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, MD, Ufuk University
Other Study IDs: 12024861-19
Record Dates: First submitted 2025-09-09; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia; PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
MeSH Terms: conditions — Fibromyalgia; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective was to determine the prevalence of fibromyalgia in women with PCOS and to examine the relationship between fibromyalgia and psychological status (depression and anxiety). Secondary objectives were to explore the potential link between fibromyalgia and insulin resistance, taking into account phenotypic differences. To assess the relationship between fibromyalgia severity and quality of life and pressure pain threshold measurements. To analyze the impact of pain and mood disorders on PCOS phenotypes and to demonstrate the role of insulin resistance in predicting fibromyalgia.

Participants will be women aged 18-40 diagnosed with PCOS according to the Rotterdam criteria, and a healthy control group of a similar age. When making a PCOS diagnosis, clinical (hirsutism, acne, menstrual irregularity), biochemical (free testosterone, DHEAS, androstenedione, etc.), and ultrasonographic (polycystic ovary morphology) findings will be evaluated. The control group will consist of healthy volunteers presenting with gynecological complaints other than PCOS and without chronic diseases.

Examination and Assessment Process Obstetrics and Gynecology Outpatient Clinic: PCOS diagnosis, demographic data, biochemical tests (glucose, insulin, HOMA-IR, etc.), and phenotyping.

Physical Therapy and Rehabilitation: Application of the 2016 ACR fibromyalgia criteria in a single-blind trial, including measurement of pressure pain threshold (algometer), fibromyalgia severity scale, and recording of Fibromyalgia Impact Questionnaire scores.

Psychological Assessment The HADS (Hospital Anxiety and Depression Scale) will be administered to assess depression and anxiety levels.

Scores obtained will be compared with fibromyalgia diagnosis and PCOS phenotypes to examine the influence of psychological factors on pain perception.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-40
2. Those diagnosed with Polycystic Ovary Syndrome by a Gynecologist and Obstetrician (according to the Rotterdam Criteria)
3. Those who agreed to participate in the study and signed the informed consent form

Exclusion Criteria:

1. Patients with underlying uterine or adnexal pathologies (endometrial polyps, adenomyosis, uterine fibroids, adnexal masses, etc.) identified by ultrasound
2. Patients with previous pelvic surgery
3. Secondary causes of hirsutism and oligomenorrhea (non-classical congenital adrenal hyperplasia, Cushing's syndrome, hypothyroidism, prolactinoma, androgen-synthesizing tumor)
4. Pregnant women
5. Patients with a history of muscular or rheumatological diseases
6. Patients with uncontrolled diabetes
7. Patients with severe psychiatric illnesses or a history of psychiatric medication/substance abuse

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients
Study Population: Participants will consist of women aged 18-40 years, diagnosed with PCOS according to the Rotterdam criteria, and a healthy control group in a similar age range.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
HADS (Hospital Anxiety and Depression Scale) | 1 month
  The HADS (Hospital Anxiety and Depression Scale) will be administered to determine depression and anxiety levels. The HADS consists of 14 questions that score both anxiety (HADS-A) and depression (HADS-D) symptoms on a scale of 0 to 3. The scores obtained will shed light on the participant's psychological state and allow for the psychological evaluation of the relationship between fibromyalgia and PCOS.
2016 ACR Fibromyalgia Criteria-The Widespread Pain Index (WPI) | 1 month
  The assessment of the WPI involves indicating persistent pain over the past seven days across five anatomical regions (upper left, upper right, lower left, lower right, axial) and 19 specific body areas (both jaws, shoulders, upper arms, lower arms, hips, upper legs, lower legs, neck, upper back, lower back, chest, and abdomen). Each region is assigned one point. The cumulative score varies from 0 to 19. 15 For a diagnosis of widespread pain, pain must be evident in a minimum of 4 out of 5 anatomical regions.
2016 ACR Fibromyalgia Criteria-Symptom Severity Scale (SSS) | 1 month
  The SSS evaluation comprises two components. In the initial section, patients evaluate the intensity of their fatigue, unrefreshing awakenings, and cognitive problems from the past week on a scale of 0 to 3. In the subsequent section, patients evaluate symptoms of headache, lower abdomen pain or cramping, and depression experienced over the preceding six months (0=none, 1=yes). The cumulative score varies from 0 to 12.
2016 ACR Fibromyalgia Criteria-The Fibromyalgia Severity Scale (FSS) | 1 month
  The Fibromyalgia Severity Scale (FSS) assessment involves the collection of WPI and SSS scores. The cumulative score varies between 12 and 31. A higher score signifies a greater disease severity. A total score exceeding 12 is required for a fibromyalgia diagnosis. A WPI of 7 or greater and an SSS score of 5 or above, or a WPI between 4 and 6 with an SSS score of 9 or above, indicate a diagnosis of fibromyalgia.
Fibromyalgia Impact Questionnaire Revised (FIQ-R) | 1 month
  It is a questionnaire designed to assess functional limitations and disabilities resulting from fibromyalgia. The questionnaire comprises a total of 21 questions divided into three sections: function, overall impact, and symptoms. Responses to each inquiry are indicated on a scale ranging from 0 to 10. The overall score is determined by summing the results: the score of the first section is divided by three, the score of the second section by one, and the score of the third section by two. Elevated scores signify a greater fibromyalgia-associated impairment.
Pressure Pain Threshold (BPT) Measurement (Algometer) | 1 month
  Pressure Pain Threshold (BPT) Measurement (Algometer): For objective pain assessment, a digital algometer will be used to measure the pressure pain threshold (the pressure level at which the patient first feels pain) at the most sensitive point on the upper trapezius muscle. The measurement will be repeated three times, and the average will be recorded.
VAS (Visual Analog Scale) | 1 month
  VAS (Visual Analog Scale): Participants will mark the intensity of their perceived pain on a 10-cm scale, rated from 0 (no pain) to 10 (unbearable pain). This method is a simple and effective way to measure a patient's subjective perception of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Elzem Bolkan Günaydın, Principal Investigator — Ufuk University
Locations (1):
- Ufuk University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided